CLINICAL TRIAL: NCT03379558
Title: Praluent® (Alirocumab) Pregnancy Exposure Registry: An OTIS Pregnancy Surveillance Study
Status: Terminated | Type: Observational
Why Stopped: (due to change in the post-marketing requirement to assess alirocumab during pregnancy)
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS14703; U1111-1195-6468 (Other: UTN)
Expanded Access: Available
Record Dates: First submitted 2017-12-15; First posted 2017-12-20 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1 : alirocumab exposed: Pregnant women diagnosed with primary hypercholesterolemia and atherosclerotic cardiovascular disease, or primary hypercholesterolemia associated with familial hypercholesterolemia and exposed to alirocumab during the current pregnancy.
  Interventions: Drug: ALIROCUMAB SAR236553 (REGN727)
- Cohort 2 : disease matched comparison: Pregnant women diagnosed of primary hypercholesterolemia and atherosclerotic cardiovascular disease, or primary hypercholesterolemia associated with familial hypercholesterolemia and unexposed to alirocumab during the current pregnancy.
- Cohort 3 : non disease comparison: Healthy pregnant women who do not have a known diagnosis of primary hypercholesterolemia and atherosclerotic cardiovascular disease, or primary hypercholesterolemia associated with familial hypercholesterolemia and have no known exposure to a known human teratogen.

INTERVENTIONS:
Drug: ALIROCUMAB SAR236553 (REGN727) — Pharmaceutical form:as per routine practice Route of administration: subcutaneous
  Other Names: Praluent®
  Groups: Cohort 1 : alirocumab exposed

SUMMARY:
Primary Objective:

To estimate the overall combined rate of major structural birth defects in infants of mothers with atherosclerotic cardiovascular disease (ASCVD) and/or familial hypercholesterolemia (FH) exposed to Praluent® (alirocumab) during pregnancy when used to treat hypercholesterolemia and to compare that rate to unexposed disease-matched and unexposed non-diseased comparison pregnancies.

Secondary Objectives:

* Secondary objectives are to estimate the rates of the outcomes in pregnancies/infants of mothers with atherosclerotic cardiovascular disease and/or familial hypercholesterolemia exposed to alirocumab during pregnancy when used to treat hypercholesterolemia and to compare that rate to unexposed disease-matched and non-diseased comparison pregnancies, and secondarily to compare the rates of these outcomes in the unexposed disease-matched pregnancies to the rates in the unexposed non-diseased comparison pregnancies.
* Safety and tolerability of alirocumab.

ELIGIBILITY:
Inclusion criteria:

Cohort 1: Alirocumab-Exposed:

Currently pregnant - Diagnosed with primary hypercholesterolemia and atherosclerotic cardiovascular disease, or primary hypercholesterolemia associated with familial hypercholesterolemia - Exposed to alirocumab for any number of days, at any dose, and at any time from the first day of the last menstrual period up to and including the end of pregnancy - Agree to the conditions and requirements of the study and provide informed consent.

Cohort 2: Disease-Matched Comparison:

Currently pregnant - Diagnosed with primary hypercholesterolemia and atherosclerotic cardiovascular disease, or primary hypercholesterolemia associated with familial hypercholesterolemia - Unexposed to alirocumab or any biologic medication during pregnancy or any time within 10 weeks prior to the first day of the last menstrual period - Agree to the conditions and requirements of the study and provide informed consent.

Cohort 3: Non-Diseased Comparison:

Currently pregnant - Not diagnosed with primary hypercholesterolemia and atherosclerotic cardiovascular disease, or primary hypercholesterolemia associated with familial hypercholesterolemia - Unexposed to alirocumab or any biologic any time in pregnancy or within 10 weeks prior to the first day of the last menstrual period - Unexposed to any known human teratogens as determined by the Organization of Teratology Information Specialists Research Center - Agree to the conditions and requirements of the study and provide informed consent.

Exclusion criteria:

Cohort 1: Alirocumab-Exposed:

First contact the Registry after prenatal diagnosis of a major structural birth defect - Enrollment in this pregnancy registry study with a previous pregnancy - Pregnancy outcome is reported retrospectively.

Cohort 2: Disease-Matched Comparison:

First contact the Registry after prenatal diagnosis of a major structural birth defect - Exposure to any alirocumab or other biologic medication during pregnancy or within 10 weeks prior to the first day of the last menstrual period - Enrollment in this pregnancy registry study with a previous pregnancy - Pregnancy outcome is reported retrospectively.

Cohort 3: Non-Diseased Comparison:

First contact the Registry after prenatal diagnosis of a major structural birth defect - Exposure to alirocumab or other biologic medication during pregnancy or within 10 weeks prior to the first day of the last menstrual period - Exposure to a known human teratogen as determined by the Organization of Teratology Information Specialists Research Center - Enrollment in this pregnancy registry study with a previous pregnancy - Pregnancy outcome is reported retrospectively.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women who enroll in the study will participate for the duration of that pregnancy.Those who deliver at least one live born infant and the infants will participate for 5 years after delivery of that infant.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-09-04 (Actual)

PRIMARY OUTCOMES:
Rate of major structural birth defects | Up to 1 year of age of the infant
  Overall combined rate of major structural birth defects in infants born to females with atherosclerotic cardiovascular disease (ASCVD) and/or familial hypercholesterolemia (FH) exposed to Praluent (alirocumab)

SECONDARY OUTCOMES:
Pregnancy outcome: Spontaneous abortion | Date of conception to 20 weeks gestation
  Rate of spontaneous abortion
Pregnancy outcome: Elective abortion | Date of conception to 20 weeks gestation
  Rate of elective abortion
Pregnancy outcome: Still birth | At birth
  Rate of still birth
Pregnancy outcome: Preterm delivery | Live birth prior to 37 weeks gestation
  Rate of preterm delivery
Infant outcome: Pattern of minor structural birth defects | Up to 1 year of age of the infant
  Specific pattern of 3 or more minor structural defects in live born infants receiving the exam
Infant outcome: Small for gestational age | At birth
  Proportion of infants who are small for gestational age on weight, length, or head circumference
Infant outcome: Postnatal growth deficiency | Up to 1 year of age of the infant
  Proportion of infants less than or equal to the 10th percentile for sex and age on weight, length, or head circumference at 1 year postnatal evaluation
Infant outcome: serious infections or hospitalizations, adverse reactions to childhood vaccinations | Up to 5 years of age of the child
  Proportion of infants who experienced serious infections or hospitalizations, and adverse reactions to childhood vaccinations
Infant outcome: adequacy of immune response | Up to 5 years of age of the child
  Proportion of infants who has adequate immune response as measured by IgG-Tetanus antibody
Infant outcome: adverse neurodevelopment | Up to 5 years of age of the child
  Proportion of infants who experienced adverse neurodevelopment
Breastfeeding/Lactation outcome | Up to 6 weeks of age of the infant
  Proportion of patients breastfeeding in the first 6 weeks after delivery
Breastfeeding/Lactation outcome | Up to 2 years of age of the child
  Proportion of patients breastfeeding exclusively for more than 2 weeks
Adverse events | Up to 5 years follow-up period
  Proportion of patients who experienced adverse events (AEs), AEs of special interest, and serious AEs

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational site UNITED STATES, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No